CLINICAL TRIAL: NCT06745986
Title: Ultrasound-Guided Fascia Iliaca Compartmental Block Versus Spinal Anesthesia in Femoral Thrombectomy: a Randomized Double-Blind Study
Brief Title: Ultrasound-Guided Fascia Iliaca Compartmental Block Versus Spinal Anesthesia in Femoral Thrombectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Port Said University hospital (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, Lecturer of anaesthesiai ntensivecare and pain managment, Port Said University hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS/17.10.109
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Fascia Iliaca Compartmental Block; Femoral Thrombectomy; Spinal Anesthesia
Keywords: Visual Analogue Score; UltraSound Guided; Fascia Iliaca Compartmental Block,; Spinal Anesthesia,; Femoral Thrombectomy
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Eighty-four cases were scheduled for femoral thrombectomy and classified into tw0 equal groups (n=42 each), spinal group received spinal anesthesia with 0.5% hyperbaric bupivacaine in a total volume in a total volume 2.5ml and fascia iliaca group received ultrasound guided fascia iliaca block with 40ml of 0.25% bupivacaine for each block. Data collected for each block were onset and duration of sensory and motor block, visual analogue scale, analgesic duration and analgesic consumption, hemodynamics and complications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fascia iliaca group (Active Comparator): The ultrasound-guided fascia iliaca compartment block (FICB) group included 42 patients who had a fascia iliaca compartment block by bupivacaine 0.25% in a total volume of 40 ml.
  Interventions: Drug: ultrasound guided fascia iliaca compartment block ( bupivacaine 0.25% )
- spinal anesthesia (Active Comparator): spinal anesthesia included 42 patients had spinal anesthesia with 2.5 ml bupivacaine 0.5%.
  Interventions: Drug: Spinal Anesthesia (bupivacaine)

INTERVENTIONS:
Drug: ultrasound guided fascia iliaca compartment block ( bupivacaine 0.25% ) — Fascia iliaca compartment block by bupivacaine 0.25% in a total volume of 40 ml.
  Arms: Fascia iliaca group
Drug: Spinal Anesthesia (bupivacaine) — spinal anesthesia by 2.5 ml bupivacaine 0.5%
  Arms: spinal anesthesia

SUMMARY:
This study aims to assess the efficiency of Fascia Iliaca Compartmental Block in patients undergoing femoral thrombectomy versus spinal anesthesia.

DETAILED DESCRIPTION:
Anesthesia for lower limb revascularization consists of general anesthesia, neuraxial anesthesia and peripheral regional block. Fascia iliaca compartment block (FICB) is an anterior approach to the lumbar plexus and it blocks femoral nerve, LFCN, and limited numbers of nearby nerves such as ilioinguinal, genitor femoral.

ELIGIBILITY:
Inclusion Criteria:

* scheduled femoral thrombectomy,
* both sexes,
* aged between 40-65 years,
* American Society of Anesthesiologists (ASA) II-III. Patients Criteria:

Exclusion Criteria:

* ASA status Grade IV, patient
* refused to participate,
* patients with contraindications to neuraxial anesthesia, such as systemic infection or history of allergy to anesthetic drugs
* infection at the site of injection.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
pain score postoperative | 24 hours
  visual analogue score (VAS), with a scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hosbital, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available upon publication of the study results in a peer-reviewed journal.
Access Criteria: Researchers and healthcare professionals conducting methodologically sound and ethically approved research